CLINICAL TRIAL: NCT06213571
Title: RISE: Remote Intervention for Strength Training in Endometrial Cancer
Brief Title: Remote Home-Based Exercise Program for Strength Training in Endometrial Cancer Survivors in Rural Areas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-008883; NCI-2023-11096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-008883 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 2 Endometrial Endometrioid Adenocarcinoma; Stage IA Uterine Corpus Cancer AJCC v8; Stage IB Uterine Corpus Cancer AJCC v8
MeSH Terms: interventions — Health Promotion; Educational Status; Interviews as Topic; Exercise Test; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (home-based exercise program) (Experimental): Participants participate in a home-based exercise program with an exercise prescription that will include resistance band and body weight exercises targeting the 5 major large muscle groups along with 3 booklets about exercise and exercise training and attend weekly exercise coaching sessions to report on exercise adherence and to progress exercise over 10 weeks on study.
  Interventions: Other: Exercise Counseling; Other: Exercise Intervention; Other: Health Promotion and Education; Other: Interview; Other: Physical Performance Testing; Other: Questionnaire Administration; Other: Telemedicine

INTERVENTIONS:
Other: Exercise Counseling — Participate in exercise coaching sessions
Other: Exercise Intervention — Participate in home-based exercise program
Other: Health Promotion and Education — Receive resistance band and exercise booklets
Other: Interview — Ancillary studies
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies
Other: Telemedicine — Participate in sessions remotely
  Other Names: Telehealth

SUMMARY:
This clinical trial studies how well a remotely delivered home-based exercise program for strength training works to positively impact endometrial cancer (EC) survivorship for patients with decreased cancer survivorship access. Cancer survivors in rural areas face barriers to supportive care, including geographic and environmental barriers to exercise and technology. Rural areas in the Midwest are underserved in terms of cancer care thus, it is essential to develop and test interventions that are scalable and can reach many individuals including those living in rural areas. Remotely-delivered exercise intervention approach allows for cancer survivors who may live far away from their primary treatment center to engage in supportive therapy via exercise interventions delivered in a sustainable context. In addition, historically black, hispanic and native endometrial cancer survivors have shorter survival and less access to survivorship care, so alternative models for healthcare delivery are needed in this underserved group. Information gained from this research may help determine whether utilizing a remotely delivered exercise program can positively impact EC survivorship for patients with decreased cancer survivorship access.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop and tailor a fully remote home-based exercise intervention for EC patients.

II. To test the recruitment and retention and acceptability of a fully remote home-based telehealth exercise intervention in older adult patients that live in rural America and are survivors of early stage, low risk endometrial cancer.

III. To measure the effectiveness of exercise intervention on quality of life in endometrial cancer patients, specifically in the realm of physical functioning.

OUTLINE:

Participants participate in a home-based exercise program with an exercise prescription that will include resistance band and body weight exercises targeting the 5 major large muscle groups along with 3 booklets about exercise and exercise training and attend weekly exercise coaching sessions to report on exercise adherence and to progress exercise over 10 weeks on study.

After completion of study intervention, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 50+
* Stage IA-IB endometrial cancer
* Grade 1-2 disease
* No recurrence documented
* Internet access
* Access to a remote device with a camera such as a computer, smartphone or tablet
* > 1 year but less than 5 years from surgery
* Primary residence in rural-urban commuting area (RUCA) (rural-urban commuting area) codes 4.0 through 10.0 or of American Indian, Alaskan Native, Black or Hispanic background

Exclusion Criteria:

* Paraplegia/hemiplegia
* No English speaking

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Retention of participants | Up to 6 months
  Assessed by the number of patients who complete 75% or more of the twice weekly exercise program.
Satisfaction with program - self-reported | 10 weeks
  Assessed by a simple participant satisfaction survey after completion of the 10-week exercise intervention. Qualitative interviews will be performed at the completion of the program regardless of level of participation to assess facilitators, barriers, and motivators to participation.
Feasibility of intervention | Up to 6 months
  Technological questions and problems that arise during the exercise intervention will be recorded to assess the ability to fully perform telehealth exercise interventions in a rural cancer population

SECONDARY OUTCOMES:
Change in physical function | Baseline; 10 weeks (end of exercise intervention); 6 months
  Assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 6b assessment, a 6-item questionnaire answered on a scale from 5 (Without any difficulty or Not at all) to 0 (Unable to do or Cannot do).

CONTACTS AND LOCATIONS:
Overall Officials: Amanika A Kumar, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials